CLINICAL TRIAL: NCT00571285
Title: Clinical Effects of Vitamin D Repletion in Patients With Parkinson's Disease
Acronym: VIDIP PILOT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marian L. Evatt, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00004539; VIDIP PILOT (Other: Other)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Nutrition; Vitamin supplement; Motor function; Non-motor function
MeSH Terms: conditions — Parkinson Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule once a week and 600 IU vitamin D daily for 26 weeks
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Placebo
- Vitamin D (Experimental): 50K IU vitamin D3 (high dose) weekly plus 600 IU Vitamin D3 capsule daily for 26 weeks
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Vitamin D3 - high dose

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 600 IU Vitamin D3 capsule daily
  Other Names: Cholecalciferol
Dietary Supplement: Vitamin D3 - high dose — 50,000 IU Vitamin D3 capsule once a week
  Other Names: Cholecalciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo capsule given once a week
  Arms: Placebo

SUMMARY:
Retrospective review of records in the Emory Movement Disorders clinic suggests vitamin D deficiency occurs in over 80% of patients with Parkinson's Disease (PD), much more frequently than in internal medicine clinics. Laboratory studies have suggested vitamin D could play a role in the development of PD. In addition, low vitamin D levels have been associated with slower walking speeds, worse memory and thinking, and depression.

DETAILED DESCRIPTION:
Retrospective review of records in the Emory Movement Disorders clinic suggests vitamin D deficiency occurs in over 80% of patients with Parkinson's Disease (PD), much more frequently than in internal medicine clinics. Laboratory studies have suggested vitamin D could play a role in the development of PD. In addition, low vitamin D levels have been associated with slower walking speeds, worse memory and thinking, and depression.

About 150 persons who have PD and low vitamin D levels will participate in this study. Subjects will be randomly (like flipping a coin) assigned to either high dose vitamin D supplement (54,200 IU weekly) or the Recommended Daily Allowance (RDA) for older persons (4200 IU weekly of vitamin D). Subjects will be examined in the clinic before, then 3- and 6- months after taking vitamin D supplement. Tests of walking speed, Parkinson's rating scales, memory tests and questionnaires of mood, anxiety and fatigue will be administered.

If this study confirms that vitamin D deficiency occurs in 80% of patients, other patients may benefit because awareness of the problem will be increased. Also, this study will help determine whether vitamin D improves patients' functioning.

Currently, there is no "standard of care" for persons with low vitamin D. At the VA Medical Center, providers use a variety of supplement regimens. The Institute of Medicine (IOM) has published 600 IU per day (4200 IU per week) as the Recommended Daily Allowance (RDA). By definition, the RDA is the amount of a vitamin or supplement that will prevent 97-98% of the population from becoming deficient.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must be able to provide informed consent or have a legal representative (defined by Georgia Law) who can give consent.
* Diagnosis of IPD, based on history of 2/3 cardinal features of PD (tremor, bradykinesia and rigidity) and definite response to dopaminergic therapy.
* Previous serum 25-OH vitamin D concentration measured by treating physician within previous 3 months.
* Eligible participants must be able to complete the study questionnaires and assessments (e.g., participant must be judged able to complete TUG at screening/baseline).
* Participants must be free of active cancer or other serious medical condition which might reasonably preclude their completing the 6-month intervention.
* Participants must be able to complete an 8 meter walk at screening evaluation.

Exclusion Criteria:

* Patients with PD, H&Y stage I-IV will be eligible to participate in this study.
* Participants must be ages 18-89 years.
* Patient with a history of hypercalcemia, hypercalciuria, liver failure, end-stage renal disease (National Kidney Foundation Classification Stage 5) or kidney stones within the past 5 years will be excluded.
* Specifically, potential participants with GFR (estimated or measured) <15 ml/min are excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visit to 3 month (Treatment Visit #1) in the TUG, timed walking task (8-meters) and UPDRS III subscore | 6 months

SECONDARY OUTCOMES:
Change from Baseline Visit to 3 month (Visit #1) and 6 month (Visit #2) in the UPDRS II, BAI-II and BDI-II score. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marian L Evatt, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States